CLINICAL TRIAL: NCT05924074
Title: Ferroptosis Study in SF3B1-mutant Myelodysplastic Syndromes (FerMDS)
Acronym: FerMDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2022/43
Record Dates: First submitted 2023-06-07; First posted 2023-06-29 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Myelodysplastic Syndromes; Ferroptosis
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SF3B1 mutant Myelodysplastic syndromes patients (MDS) (Experimental): Patients diagnosed with MDS carrying the SF3B1 somatic mutation associated myelodysplastic neoplasm with ring sideroblasts
  Interventions: Biological: Biological sampling
- Monoclonal Gammapathy of Unknown Significance patients (MGUS) (Active Comparator): MGUS patients, referred to as normal bone marrow controls
  Interventions: Biological: Biological sampling

INTERVENTIONS:
Biological: Biological sampling — The procedure will consist of an additional bone marrow sample and blood sample

SUMMARY:
Myelodysplastic syndromes (MDS) are clonal diseases of hematopoietic stem cells (HSC) characterized by dysplastic and inefficient hematopoiesis related to excessive progenitor cell death. Ferroptosis is a recently described cell death mechanism and we think that it could be a major player in the pathophysiology of MDS, involved in the cell death that characterizes these diseases and contributing to cytopenias. The study aims to demonstrate that there is a significant activation of this phenomenon in MDS patients compared to a population of subjects without MDS.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are hematological malignancies characterized by a defect in blood cells production. Their pathophysiology remains poorly understood, but an excessive death of progenitor cells is considered as a key mechanism contributing to the appearance of cytopenia. Furthermore, it is known that there are abnormalities of iron metabolism in MDS, especially in patients with ring sideroblasts and SF3B1 mutation. The classical therapeutic strategy in MDS relies on symptomatic management of cytopenias (transfusions, growth factors) associated with demethylating agents in high-risk forms. Unfortunately, these treatments only stabilize the disease and only allogeneic bone marrow transplantation (reserved to limited number of patients) can cure the patients. Therefore, there is a urgent need to identify new therapeutic targets in these diseases.

An excessive apoptosis activation has been shown in MDS for a long time. However, other cell death pathways could also contribute to their pathophysiology. Among them, ferroptosis, a cell death process triggered by the accumulation of free iron in the cell, seems to be a promising candidate.

The project is proposed to study ferroptosis in SF3B1-mutant MDS patients. An additionnal bone marrow sample will be aspirate at diagnosis. Ferroptosis will be analyzed using flow cytometry (labeling of peroxidized lipids with C11-BODIPY). The percentage of cells in ferroptosis will be compared between SF3B1-mutant MDS patients and control patients (patients evaluated for Monoclonal Gammapathy of Unknown Significance-MGUS). The presence of an excess of ferroptosis in SF3B1-mutant MDS patients will be correlated to clinico-biological parameters. No follow up will be be performed.

ELIGIBILITY:
Inclusion Criteria:

For all :

* Patients of legal age (age ≥ 18 years)
* Subjects affiliated to or benefiting from a social security scheme
* Free, written and informed consent signed by the participant and the investigator

For MDS patients :

* Sampling at diagnosis for MDS patients (WHO 2016 criteria)
* Presence of ring sideroblasts on bone marrow smear

For MGUS patients :

- Sampling as part of the exploration of monoclonal gammopathy of undetermined significance (MGUS) for controls (WHO 2016 criteria).

Exclusion Criteria:

For all

* Patient transfused with red blood cells within 120 days prior to collection
* Patients treated with haematopoietic growth factors (EPO, TPO, G-CSF) within 30 days prior to collection
* Patients with conditions that affect systemic iron metabolism: hemochromatosis, Gaucher disease, ferroportin disease, porphyria cutanea tarda
* Person under a legal protection measure (legal protection, guardianship or curatorship)
* Person deprived of liberty by judicial or administrative decision
* Person who is unable to give consent
* Subject who is in an exclusion period after another study or who has participated in another interventional drug study within 30 days prior to entry into the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of cells undergoing ferroptosis in SF3B1-mutant MDS patients compared to MGUS patients | At Baseline
  Mean values for the proportion of ferroptose cells will be compared between arms, using comparative statistical methods (Student's t test, Student's test for unequal variances or Wilcoxon test)

SECONDARY OUTCOMES:
Percentage of cells undergoing ferroptosis in the different bone marrow subpopulations (stem cells, progenitors, and erythroid and myeloid precursors at different stages of differentiation) of SF3B1-mutant MDS patients | At Baseline
  Mean values for the proportion of ferroptose cells among the different bone marrow subpopulations will be compared between arms, using comparative statistical methods (Student's t test, Student's test for unequal variances or Wilcoxon test)
Biological characteristics of SF3B1-mutant MDS patients with an excess of cells undergoing ferroptosis in the bone marrow compared to MGUS controls | At baseline
  Biological differences in number (1 to 3) and type of cytopenias (anemia, thrombocytopenia, neutropenia) in SF3B1-mutated MDS patients will be studied and statistically compared with the MGUS control group, based on the number of ferroptosis cells observed by cytometry
Clinical characteristics of SF3B1-mutant MDS patients with an excess of cells undergoing ferroptosis in the bone marrow compared to MGUS controls | Through study completion, up to 2 years
  Overall survival after diagnosis, progression-free survival (evolution of MDS towards a higher-grade hemopathy or death) in SF3B1-mutated MDS patients will be studied and statistically compared with the MGUS control group, based on the number of ferroptosis cells observed by cytometry

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Bordeaux, Laboratoire d'Hématologie, Pessac
  - CHU de Bordeaux, Service de Médecine Interne, Pessac
  - CHU de Bordeaux, Service Hématologie Clinique et Thérapie Cellulaire, Pessac

IPD SHARING:
Plan to Share IPD: No